CLINICAL TRIAL: NCT06100419
Title: Is Serratus Posterior Superior Intercostal Plane Block Effective in Modified Radical Mastectomy Surgeries?
Brief Title: SPSIP Block in Breast Surgeries for Postoperative Analgesia
Acronym: SPSIPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Fatih Balci, Specialist/Department of Anaesthesiology and Reanimation, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPSIPB
Record Dates: First submitted 2023-10-14; First posted 2023-10-25 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Postmastectomy Pain
Keywords: serratus posterior superior intercostal plane block; regional anaesthesia; postmastectomy pain; interfascial plane blocks

STUDY DESIGN:
Intervention Model Description: case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Block (Experimental): This group consists of patients who underwent SPSIP block.
  Interventions: Procedure: serratus posterior superior intercostal plane block

INTERVENTIONS:
Procedure: serratus posterior superior intercostal plane block — With this newly introduced procedure added to the literature, patients undergoing breast surgeries are expected to experience reduced pain.
  Other Names: SPSIPB

SUMMARY:
The aim of this clinical study is to demonstrate that pain following breast surgeries can be reduced through the application of serratus posterior superior intercostal plane block (SPSIPB). Seven patients scheduled for breast surgery were included in the study. The primary research question it seeks to address is as follows: • Can SPSIPB be applied to reduce pain following breast surgeries? Participants are expected to provide accurate responses to the researcher's questions for the assessment of postoperative pain.

DETAILED DESCRIPTION:
Postoperative analgesia techniques for breast surgeries encompass options such as Paravertebral Block, Erector Spinae Plane Block, Serratus Anterior Plane Block, and Pectoral Nerve Blocks. Although the Paravertebral Block is considered the gold standard for postmastectomy pain relief, its limited usage is primarily attributed to complications. SPSIPB's potential in thoracic surgeries has been noted, offering a broad sensory block suitable for MRM and axillary lymph node dissection. In this study, the effectiveness of SPSIP block for post-mastectomy pain has been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who will undergo breast surgery

Exclusion Criteria:

* unstable patients
* patients with bleeding disorders
* Patients allergic to local anesthetic drugs
* Patients who did not agree to participate in the study
* Patients with infection at the application site

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Since patients undergoing breast surgery were selected, the group consists of female patients.
Enrollment: 7 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
numeric rate scores (NRS) | first 24 hours
  The pain levels of patients are indicated with a number between 1 and 10. its means: 0=no pain, 10=worst pain.

SECONDARY OUTCOMES:
total tramadol consumption | first 24 hours
  The total analgesic quantity that patients will consume for pain reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No